CLINICAL TRIAL: NCT05897606
Title: Effect of Multi Vitamin and Mineral Supplementation of Liver Enzymes and Sonography in Patient With Non-alcoholic Fatty Disease (NAFLD); RCR
Brief Title: Effect of Multi Vitamin and Mineral Supplementation of Liver Enzymes and Sonography in Patient With NAFLD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sulaimany Polytechnic university (Other)
Responsible Party: Principal Investigator, Hawal Lateef Fateh, Dr Hawal Lateef Fateh, Sulaimany Polytechnic university
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KTC1211
Record Dates: First submitted 2023-05-24; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Minerals

STUDY DESIGN:
Intervention Model Description: Intervention group received multivitamin and minerral
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- effect multivitamin and minerals on NAFLD for 12 weeks (Experimental): The intervention group received one capsule of multivitamin and minerals supplements every day, one hour after breakfast, for 12 weeks.
  Interventions: Combination Product: Multiviamins and minerals
- Placebo (Placebo Comparator): the control group took a placebo prepared with the same shape and size of supplements.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Multiviamins and minerals — The intervention group received one capsule of multivitamin and minerals supplements every day, one hour after breakfast, for 12 weeks.
  Arms: effect multivitamin and minerals on NAFLD for 12 weeks
Combination Product: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study was performed on 160 participants, to ensure the impact of multi vitamin and mineral to reduce NAFLD

DETAILED DESCRIPTION:
This study was performed on 160 participants, to ensure the impact of multi vitamin and mineral to reduce NAFLD.

Participants were randomly selected to participate in the study. Then divided into the groups (intervention and placebo). Intervention received supplementation for 12 weeks and placebo received same capsule was made for placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants with NAFLD diagnosed

Exclusion Criteria:

* subjects who in the last 6 months received vitamin or mineral supplementation, those with chronic conditions such as diabetes, hypertension, and heart disease, unwillingness to continue the study protocol, lactating women and pregnant women.

Ages: 22 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Multivitamin and minerals supplementation has role in reduce liver enzymes | 12 weeks
  Multivitamin and minerals supplement was given for 12 weeks and has role in reduce Serum Bilirubin, alkaline phosphatase (ALP), alanine transaminase (ALT), and liver enzyme was measured by blood sampling tests.

CONTACTS AND LOCATIONS:
Overall Officials: HAWAL F Lateef, Msc, Principal Investigator — Nursing Department, Kalar Technical College, Sulaimani polytechnic university, Sulaimani, Iraq
Locations (1):
- Hawal Fateh, Kurdistan, Kalar, Iraq

IPD SHARING:
Plan to Share IPD: No